CLINICAL TRIAL: NCT03540550
Title: Modification of the Gut Microbiota Following the Consumption of Inulin-rich Vegetables: Effect on Gut Tolerance, Transit, Behaviour and Digestion in Healthy Humans
Brief Title: Effects of a Diet Based on Inulin-rich Vegetables on Gut Health and Nutritional Behaviour in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B403201627275
Record Dates: First submitted 2018-05-08; First posted 2018-05-30 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary intervention (Experimental)
  Interventions: Other: Diet based on inulin-rich vegetables

INTERVENTIONS:
Other: Diet based on inulin-rich vegetables — During two weeks, healthy subjects were instructed to adhere to a controlled diet based on ITF-rich vegetables (±15 g ITF/day).

SUMMARY:
Inulin-type fructans (ITF) are fermentable dietary fibres that can confer beneficial health effects through changes in the gut microbiota. However, their effect on gut sensitivity and nutritional behaviour is a matter of debate.

The investigators evaluated, in healthy individuals, the impact of shifting from their usual food habits towards a diet based on the daily consumption of ITF-rich vegetables on gut microbiota, gastro-intestinal symptoms and food-related behaviour.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 25 kg/m²
* Caucasian ethnicity
* Hydrogen producers (assessed by hydrogen breath test)

Exclusion Criteria:

* Smokers
* Laxative consumption (<4 weeks)
* Severe intestinal problems
* Psychiatric problems or use of antipsychotic
* Consumption of antibiotics, pro/prebiotics, fibre dietary supplement, or any molecules that modifies the intestinal transit (<6 weeks)
* Specific dietary practise (vegetarian, vegan,...)
* Specific dietary treatment (<6 weeks) (e.g. high protein diet)
* Excessive alcohol consumption (>3 glasses/day)
* Consumption of the following drugs: proton pump inhibitor, antidiabetic drugs, cholesterol lowering drugs
* Inconclusive acceptability test (regarding the protocol of the intervention and the vegetables used in the protocol)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-04-12 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition | 33 days
  Gut microbiota composition is assessed by 16S rRNA pyrosequencing. This analysis allows to obtain the relative abundance (%) of the different bacterial taxa and OTUs (operational taxonomic units).

SECONDARY OUTCOMES:
Gut microbiota fermentation in vivo | 33 days
  Gut microbiota fermentation is assessed in vivo by an hydrogen breath test. After an oral load of purified inulin, the level of expired hydrogen (ppm) is measured.
Gut microbiota fermentation in vitro | 14 days
  Gut microbiota fermentation is assessed in vitro by the measurement of total gas (ml/g of dry matter) produced from subject feces incubated with inulin-rich substrates.
Gastrointestinal Symptoms | 33 days
  Gastrointestinal symptoms were assessed by Visual Analogue Scale (horizontal line of 100 mm). Each subject completed seven separate scales, one for each symptom (rumble, burp, bloating, discomfort, nausea, flatulence, cramp), ranging from "no sensation" (0 mm) to "very severe sensation" (100 mm).
Appetite-related feelings | 33 days
  Appetite-related feelings were assessed by Visual Analogue Scale (horizontal line of 100 mm). Each subject completed seven separate scales, one for each appetite-related feeling (satiety, intention to eat, fullness, sweet envy, very sweet envy, fat envy, salt envy), ranging from "no sensation" (0 mm or 100 mm depending on the feeling) , to "very strong sensation" (0 mm or 100 mm depending on the feeling).
Correlation of gastrointestinal symptoms with gut bacteria | 33 days
  The levels of gastrointestinal symptoms were correlated (Spearman correlations) with the relative abundance of bacterial taxa and OTUs (operational taxonomic units)
Short chain fatty acids production | 14 days
  Short chain fatty acids (SCFAs) production was assessed in vitro by the measurement of total SCFAs (mg/g of dry matter) produced from subject feces incubated with inulin-rich substrates.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Thissen, Pr., Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hiel S, Bindels LB, Pachikian BD, Kalala G, Broers V, Zamariola G, Chang BPI, Kambashi B, Rodriguez J, Cani PD, Neyrinck AM, Thissen JP, Luminet O, Bindelle J, Delzenne NM. Effects of a diet based on inulin-rich vegetables on gut health and nutritional behavior in healthy humans. Am J Clin Nutr. 2019 Jun 1;109(6):1683-1695. doi: 10.1093/ajcn/nqz001. PMID 31108510